CLINICAL TRIAL: NCT02857439
Title: Creating a Diagnostic Decision Rule for Shoulder Injury: CASH-trial
Acronym: CASH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zaans Medisch Centrum (Other)
Responsible Party: Principal Investigator, K. Rijsbergen, Research intern, Zaans Medisch Centrum
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CASH Zaansmc
Record Dates: First submitted 2016-07-29; First posted 2016-08-05 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-08

CONDITIONS: Trauma
Keywords: Trauma of the shoulder
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MD as first examiner (Other): Patients will be examined according to a standardized physical examination item list
  Interventions: Other: Standard diagnostic item list
- Triage nurse as first examiner (Other): Patients will be examined according to a standardized physical examination item list
  Interventions: Other: Standard diagnostic item list

INTERVENTIONS:
Other: Standard diagnostic item list — All consecutive patients are assessed by both examiners, according to a standardized physical examination item list.

SUMMARY:
What combination of ≤ 6 clinical variables will give the highest specificity for indicating significant shoulder injuries (fractures or dislocations) with a set sensitivity of ≥ 97%?

Although shoulder trauma is a common injury, there is no clinical decision rule to determine the necessity for radiography for these traumas. With this trial the investigators aim to develop such a rule to reduce the amount of radiographs without missing any significant injuries.

The primary objective is to compose a set of clinical diagnostic criteria predictive of shoulder fractures or dislocations that would reduce the amount of radiographs without missing any significant injuries. A second objective is to determine if the clinical decision rule is applicable for triage use.

DETAILED DESCRIPTION:
The CASH (Clavicle-AC-Joint-Sub-capital-Humerus) trial is designed as a cross sectional interobserver study. It will randomize between first examiner of the patient to determine applicability for triage use and use a list of 19 criteria to determine a clinical decision rule for significant shoulder injuries.

Method/intervention After admittance to the ED, all consecutive shoulder injury patients will be assessed for eligibility in the study. After informed consent is given, the patient will be randomized for first observer (ED physician or triage nurse) to be examined, which means they will be assessed in duplo.

The patient will be examined by means of a score form, which contains 19 different diagnostic criteria. The criteria are grouped: anamnesis, inspection, palpation and pain/range of motion(ROM). After completing the list, patients will get a full set of shoulder x-rays: shoulder AP- and axial-view, and clavicle AP and 30' cranio-caudal view.

The trial participation for the patient will be completed at this point and final diagnosis and treatment are provided by the ED physician according to his/her own findings and interpretation of the radiographs. For the study, the radiographs will be reassessed by one consultant radiologist specialized in skeletal trauma.

ELIGIBILITY:
Inclusion Criteria:

* Aged18-65 years
* Trauma <48h

Exclusion Criteria:

* Any prior ipsilateral shoulder surgery.
* Any diseases of the bones potentially influencing fracturability (osteogenesis imperfecta, osteoporosis, achondroplasia, M. Kahler, chronic (> 1yr) prednisone use > 5mg)
* Any shoulder injury as part of a multi-trauma or high energy trauma (HET) with distractible injuries
* Any condition that will influence the perception of pain (e.g. alcohol intoxication, psychiatric problems, mental retardation)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy (sensitivity and specificity) of the clinical variables assessed with the score form. | An average of 12 to 18 months

SECONDARY OUTCOMES:
Interobserver agreement for each clinical variable between both observers determined with the Cohen's kappa coefficient | An average of 12 to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Kim Rijsbergen, BSc, Principal Investigator; Robert Jan Derksen, MD, Study Director — Zaans Medisch Centrum
Locations (1):
- Zaans Medisch Centrum, Zaandam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Stiell IG, Greenberg GH, McKnight RD, Nair RC, McDowell I, Worthington JR. A study to develop clinical decision rules for the use of radiography in acute ankle injuries. Ann Emerg Med. 1992 Apr;21(4):384-90. doi: 10.1016/s0196-0644(05)82656-3. PMID 1554175
- [Background] Bachmann LM, Kolb E, Koller MT, Steurer J, ter Riet G. Accuracy of Ottawa ankle rules to exclude fractures of the ankle and mid-foot: systematic review. BMJ. 2003 Feb 22;326(7386):417. doi: 10.1136/bmj.326.7386.417. PMID 12595378
- [Background] Stiell I, Wells G, Laupacis A, Brison R, Verbeek R, Vandemheen K, Naylor CD. Multicentre trial to introduce the Ottawa ankle rules for use of radiography in acute ankle injuries. Multicentre Ankle Rule Study Group. BMJ. 1995 Sep 2;311(7005):594-7. doi: 10.1136/bmj.311.7005.594. PMID 7663253